CLINICAL TRIAL: NCT00665327
Title: A Study of Avelox for Treatment of Elderly Patients With Community Acquired Pneumonia
Brief Title: Avelox for Treatment of Elderly Patients With Community Acquired Pneumonia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10872
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Pneumonia
Keywords: Community Acquired Pneumonia; Pneumonia,; CAP
MeSH Terms: conditions — Pneumonia; Community-Acquired Pneumonia | interventions — Moxifloxacin; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Avelox (Moxifloxacin, BAY12-8039)
- Arm 2 (Active Comparator)
  Interventions: Drug: Levofloxacin

INTERVENTIONS:
Drug: Avelox (Moxifloxacin, BAY12-8039) — Moxifloxacin 400 mg IV QD for a minimum of two doses followed by moxifloxacin 400 mg PO QD for a total treatment duration of 7 to 14 days
  Arms: Arm 1
Drug: Levofloxacin — Levofloxacin 500 mg IV QD for a minimum of two doses followed by Levofloxacin 500 mg PO QD for a total treatment duration of 7 to 14 days. For patients who have a documented or calculated creatinine clearance of 20 - 49 ml/minute, the IV and PO dose of Levofloxacin will be a 500 mg loading dose followed by 250 mg QD for a total treatment duration of 7 to 14 days
  Arms: Arm 2

SUMMARY:
This study was to assess the safety of sequential intravenous (IV)/oral (PO) moxifloxacin (Avelox®) compared with sequential IV/PO levofloxacin (Levaquin®) in the treatment of elderly subjects (aged ≥ 65 years) with community-acquired pneumonia (CAP) who required initial IV therapy. This study also included an assessment of the clinical and bacteriologic effectiveness of both drugs.

ELIGIBILITY:
Inclusion Criteria:

* Presence of radiological evidence of a new or progressive infiltrate(s) consistent with bacterial pneumonia and at least 2 of the following:
* Productive cough with purulent or mucopurulent sputum/tracheobronchial secretions or change in the character of sputum (increased volume or purulence)
* Dyspnea or tachypnea
* Rigors or chills- Pleuritic chest pain
* Auscultatory findings on pulmonary examination of rales/crackles and/or evidence of pulmonary consolidation- Fever or hypothermia
* White blood cell count >/= 10000/mm3 or >/= 15% immature neutrophils, regardless of the peripheral WBC count, or leukopenia with total WBC count < 4500/mm3

Exclusion Criteria:

* Known hypersensitivity to fluoroquinolones- Presence of end-organ damage or shock with need for vasopressors for > 4 hours at the time of study entry
* Need for mechanical ventilation at study entry
* Implanted cardiac defibrillator.- Significant bradycardia with heart rate < 50 beats/minute.
* Hospitalized for > 48 hours before developing pneumonia.
* Systemic antibacterial therapy for more than 24 hours within 7 days of enrollment unless the patient was deemed a treatment failure after receiving greater than 72 hours of a non-fluoroquinolone antibiotic.
* Co-existent disease considered likely to affect the outcome of the study (e.g. active lung cancer, connective tissue disease affecting the lungs, bronchiectasis).
* Mechanical endobronchial obstruction (e.g. endobronchial tumor).
* Known or suspected active tuberculosis or endemic fungal infection
* Neutropenia (neutrophil count < 1000/Microliter).
* Chronic treatment (equal or longer than 2 weeks) with known immunosuppressant therapy (including treatment with > 15 mg/day of systemic prednisone or equivalent).
* Patient with known HIV infection and a CD4 count < 200/mm3 .
* Known severe hepatic insufficiency .
* Renal impairment with a baseline measured or calculated serum creatinine clearance < 20 mL/min. If a recent value for a 24 hour creatinine clearance is not available then the creatinine clearance should be calculated using the Cockcroft-Gault formula .
* Known prolongation of the QT interval or use of Class IA or Class III antiarrhythmics (e.g., quinidine, procainamide, amiodarone, sotalol).
* Uncorrected hypokalemia.
* Previous history of tendinopathy with quinolones.
* Previously entered in this study.- Participated in any clinical investigational drug study within 4 weeks of screening.
* Known or suspected concomitant bacterial infection requiring additional systemic antibacterial treatment.
* Patients with a history of a hypersensitivity reaction to multivitamin infusion (MVI) or pre-existing hypervitaminosis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 401 (Actual)
Dates: Start 2002-11; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Incidence of a composite safety end point (including cardiac arrest, sustained and non-sustained ventricular tachycardia), based on digital Holter ECG recordings | First 72 hours of study participation

SECONDARY OUTCOMES:
Incidence of a composite safety end point (including atrial fibrillation sustained and unsustained supraventricular tachycardia, third degree AV block and long RR pauses), based on Holter | First 72 hours of study participation
Adverse Events Collection | Up to 7-14 days post-therapy
Clinical Response | Day 3-5 during treament, 7-14 days post-therapy
Mortality attributable to pneumonia | 7-14 days post-therapy
Bacteriological Response | 7-14 days post-therapy
Overall cost of hospitalization | Up to 7-14 days post-therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (68):
- United States (67):
  - Mobile, Alabama
  - Tucson, Arizona
  - Brea, California
  - Fullerton, California
  - La Jolla, California
  - Madera, California
  - Bridgeport, Connecticut
  - Farmington, Connecticut
  - Stamford, Connecticut
  - Brandon, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Austell, Georgia
  - Blue Ridge, Georgia
  - Columbus, Georgia
  - Fort Gordon, Georgia
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Coeur d'Alene, Idaho
  - Elk Grove Village, Illinois
  - Springfield, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Cumberland, Maryland
  - Kalamazoo, Michigan
  - Royal Oak, Michigan
  - Duluth, Minnesota
  - Columbia, Missouri
  - St Louis, Missouri
  - Anaconda, Montana
  - Omaha, Nebraska
  - Holmdel, New Jersey
  - Neptune City, New Jersey
  - Newark, New Jersey
  - Albany, New York
  - Johnson City, New York
  - Kingston, New York
  - Manhasset, New York
  - Mineola, New York
  - New York, New York
  - Syracuse, New York
  - Chapel Hill, North Carolina
  - Elizabeth City, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Lima, Ohio
  - Tulsa, Oklahoma
  - Allentown, Pennsylvania
  - Beaver, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Summerville, South Carolina
  - Jackson, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - El Paso, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Lynchburg, Virginia
  - Norfolk, Virginia
- San Juan, Puerto Rico